CLINICAL TRIAL: NCT06924307
Title: In-Home Parent-Child Training System: Validation Study
Brief Title: Parent-Child EF Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koronis Biomedical Technologies (Industry)
Collaborators: University of Minnesota (Other); National Institute of Mental Health (NIMH) (NIH); Mount Sinai General Pediatrics Faculty Practice (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-2024; 5R44MH121664 (NIH)
Record Dates: First submitted 2025-03-21; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Intervention to Promote Healthy Development of Executive Function (EF) Skills in Young Children
Keywords: Executive Function

STUDY DESIGN:
Intervention Model Description: The study will involve identical procedures across both sites to ensure consistency and comparability. Participating families will be randomly assigned (with stratification) to the MindMovers or active control condition, instructed to utilize the assigned app for 4 weeks, and given pre, post, and delayed post-test assessments. The primary caregiver for the purposes of the study and the child will come to the site for a pre-test visit. Caregivers will be trained to use the assigned app by a researcher. The MindMovers will include 20 activities and 2 video games. Then families will have a 4-week in-home practice period, with the goal of 20-min per day on 20 training days (5 days per week).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mind Movers Intervention (Experimental): This arm will be administered the Mind Movers Intervention
  Interventions: Device: Executive Function Intervention
- Control (No Intervention)

INTERVENTIONS:
Device: Executive Function Intervention — The intervention is an in-home cognition training system that provides parents with a modular series of short, easy-to-follow, collaborative cognitive training activities they will share with their child to address the needs of families with young children identified with deficits in executive function (EF), a critical cognitive process associated with self-control. The system employs a novel two-generational training model that views parental involvement as a critical component of the intervention process. In this model, an engaging, parent-facing smartphone application will deliver personalized daily training activities consisting of both traditional hands-on activities as well as collaborative, parent-controlled, child-facing video games. This approach supports multiple pathways for learning and building strong personal relationships between parent and child.
  Arms: Mind Movers Intervention

SUMMARY:
Koronis Biomedical Technologies Corporation (KBT) is developing a cognitive intervention to promote healthy development of Executive Function (EF) skills in young children by leveraging a smartphone-based training regime designed for parents.

DETAILED DESCRIPTION:
The proposed intervention includes non-computerized play activities, child-facing EF video games with parental controls, and a clinician-facing portal to monitor and analyze progress, building on prior feasibility studies and expanding validation with a larger sample size and additional outcome variables. EF skills provide a foundation for learning and adaptation across a wide range of situations, and are necessary for emotion regulation, social interactions, and school/work performance. Difficulties with EF skills serve as a transdiagnostic indicator of many clinical conditions with childhood onset, including ADHD, autism, and conduct disorder, among others. There have been major advances in the reliable and validated assessment of EF skills in children, such as the NIH Toolbox for the Assessment of Neurological and Behavioral Function (Zelazo et al., 2013) and the Minnesota Executive Function Scale (Carlson & Zelazo, 2014). Parents of children with potential delays in EF skills have an unmet need, however, for an affordable and timely intervention option. This research seeks to fill this need by developing an in-home cognitive training system that provides parents with short (20-minute), adaptive collaborative cognitive training activities they will engage in with their child. This study will be conducted at two sites: the University of Minnesota's Institute of Child Development (ICD) and the Mount Sinai General Pediatric Faculty Practice. Both sites provide exceptional resources and expertise in early childhood development, EF research, and parent-child interaction studies. Their complementary strengths ensure a robust foundation for participant recruitment and data collection.

Preliminary Data - In Phase I, KBT engineers, working together with researchers from the University of Minnesota, developed and tested a prototype Executive Function (EF) cognitive training system. The system employs a novel two-generational training model that views parental involvement as a critical component of the intervention process. In this model, an engaging, parent-facing smartphone/tablet application delivers personalized daily training activities consisting of both short, easy-to-follow, hands-on cognitive training activities, as well as collaborative, parent-directed, child-facing video games. In Phase I, a demonstration child-facing video game called Spin the Pots was fully developed and tested. Our approach supports multiple pathways for learning and the building of strong personal relationships between parent and child. Parents were issued the MindMovers and Spin the Pots via the Google Play store and trained over a Zoom session with the Project Coordinator. They were instructed to use the apps with their child for 10 days within a 14-day period, for a total of 20 minutes per day at any time of their choosing (7 minutes for Spin the Pots and 13 minutes for the parent-child activities). Nineteen families completed the study (95%). One family withdrew prior to the post-test due to lack of time.

Usage Data - Parents used the offline activities with their child an average of 8.06 separate days (SD=3.13, range= 2-13), totaling an average of 148.4 minutes (SD=83.9, range=14.8-325) or 141.6% the recommended per-session dose. Children played Spin the Pots an average of 5.95 separate days (SD=2.35; range=2-10), totaling an average of 54.4 minutes (just under one hour) (SD=38.7, range=12.4-144.7), or 130.6% the recommended per-session dose. This usage reflects a positive experience in busy, real-life conditions.

Quantitative Results - Participating children showed the full range of ability on the working memory game Spin the Pots. Performance (Highest Level Passed) was correlated with age, as expected, r(20) = .391, p = .088. The more times children played the game, the better they got, r(20) = .66, p = .002. Parents began each "MindMovers" activity at the lowest level (1) to help children become acquainted with the basic objective, and then advanced to higher levels to help maintain a challenge as their child improved, which is important for EF growth. There was large variability in usage of each activity across families, yet parents generally moved up the scale on each activity, ending at level 4 (out of 5) on average during the study period. Age was associated with the highest mastery level attempted (rs = .29-.40), although these were not statistically significant given the small sample size in this usability study. There were no sex differences on Spin the Pots or the Launchpad activities. Our Spin the Pots video game was significantly correlated with the "gold standard" Minnesota Executive Function Scale (after controlling for age, r-Pretest = .43, r-Posttest = .53), as well as three of the parent-child activities (BINGO, Breathing, and Freeze Dance). The MEFS was also positively related to Breathing and Freeze Dance. This study provided preliminary evidence that our tool has construct validity, although it did not result in improved EF scores in such a small sample over a brief (2-week) period. A longer time period with a larger variety of activities is needed to fully assess the impact of the training. Qualitatively, parent surveys indicated the app was easy to use and enjoyed by both children and parents.

Purpose of the study:

The purpose of the study is to expand and validate a low-cost, developmentally appropriate, smartphone-based training regimen for parents to help promote parent-child interactions that support the healthy development of EF skills in young children, including those who have been identified as having deficits in their EF skills. Specific Aims 1-4 of the project will result in a smartphone-based EF-training application that provides parents with 20 activities to instruct and support traditional non-computerized play, and two child-facing EF video games with parental controls. Aim 5 is to develop a clinician-facing administrator portal for storing, analyzing, and displaying participants' progress in using the tool and EF assessment results. The specific aim of this human subjects protocol is to assess the validity of the system when used for a longer period of time by families (Aim 6). It includes a larger sample size than the feasibility study, as well as additional outcome variables and a delayed post-test.

The study is a pre/post/delayed post-test design with two conditions including random assignment using a randomization tool (e.g., Sealed Envelope), balanced on child age and sex and parent's education level.

A total of N = 140 children aged 24 to 71 months, and their primary caregivers will be recruited to participate in the validation study. According to pilots and attrition, we anticipate a final sample size of N ≥ 50-70 at each site.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 2-5 years.
* Caregivers/guardian of the participating child.

Exclusion Criteria:

* Children with physical disabilities affecting vision, hearing, or basic mobility.
* Children with severe developmental delays or disorders
* Parents or caregivers who cannot read and understand English

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Parent Knowledge Questionaire | Week 1, 5, 9
  Understanding of EF (From Parent)
Minnesota Executive Function Scale (MEFS) | Week 1, 5, 9
  Standardized EF Assessment (From Child)
Peg Tapping | Week 1, 5, 9
  EF Assessment (From the Child)
Forward/Backward Word Span | Week 1, 5, 9
  EF Assessment (From the Child)
Behavior Rating Inventory of Executive Functioning - Preschool (BRIEF-P) | Week 1, 5, 9
  EF questionnaire (about Child from the Parent)
Self-reported usage | Week 5
  Usage of Apps (Parent)
ReadyRosie App Usage | During the intervention
  The total number of videos viewed by participants, representing overall engagement frequency with the app.
ReadyRosie Learning Outcome Opportunities | During the intervention
  The cumulative number of learning opportunities accessed by participants, categorized into four developmental domains: Language and Literacy, Math, Social-Emotional, and Health and Well-Being. This reflects both viewing activity and engagement with the child during or after the video.
ReadyRosie Family Outcome Opportunities | During the intervention
  The aggregate number of instances in which families engaged with their child in activities tagged according to the Head Start Family Engagement Framework. This measure captures the breadth of family involvement across key developmental categories.
MindMovers Usage Frequency | During the intervention
  The total number of times participants logged into the app, including timestamps that indicate the day and time of each login.
MindMovers Activity Duration | During the intervention
  The recorded time (in minutes and seconds) spent on each game or activity, as tracked by the app's internal portal.
MindMovers Game/Activity Levels Achieved | During the intervention
  Each game session records both the session duration and the final level reached. For both Spin the Pots and Beachcomber, the highest achievable level is 7. This metric captures the highest level completed by the child participant per session.
MindMovers Reflection Prompts | During the intervention
  The duration (ranging from 1 to 20 minutes) of parent-guided reflection activities conducted after gameplay. Parents and children rated their enjoyment and engagement with the activity on a 5-point scale.
MindMovers Badges Earned | During the intervention
  The total number of badges awarded to participants during gameplay in Spin the Pots and Beachcomber. Badges are earned based on in-game performance and milestones.

SECONDARY OUTCOMES:
Family Information Questionnaire | Week 1
  Family Demographics (From the Parent)
Parenting Stress Index - Short Form | Week 1, 5, 9
  Stress related to parenting (From the Parent)
Children's Social Understanding Scale - Short Form | Week 1, 5, 9
  Social understanding questionnaire (far transfer). (Collected from Parent)
Ages & Stages Questionnaires: Social-Emotional, Second Edition (ASQ:SE-2) | Week 1, 5, 9
  Social-emotional learning (Collected from the Parent)
Usability Survey | Week 5
  App usability (From Parent)
Open-ended Interview | Week 5
  Thoughts/feelings about the App (From Parent)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie M. Carlson, PhD, Principal Investigator — University of Minnesota; Blair Hammond, MD, Principal Investigator — Mount Sinai General Pediatrics
Locations (2):
- United States (2):
  - University of Minnesota, Institute of Child Development, Minneapolis, Minnesota
  - Mount Sinai General Pediatrics, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] S. M. Carlson and P. D. Zelazo, "Minnesota Executive Function Scale," Reflect. Sci. Inc St Paul MN, 2014.